CLINICAL TRIAL: NCT06986252
Title: Effect of Nurse-led Education on Health, Quality of Life and Sexual Health for Patients Undergoing Endovascular Intervention for Abdominal Aortic Aneurysm
Brief Title: Effect of Nurse-led Education on Health, Quality of Life and Sexual Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgical specialist nurses appointed to the intervention resigned from employment.
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DNR064-13
Record Dates: First submitted 2025-04-01; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Aortic Aneurysms (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): the intervention group received standard care plus they were also offered two consultations at a specialist surgical nurse-led clinic
  Interventions: Other: Consultation
- Control (No Intervention): The control group received standard care.

INTERVENTIONS:
Other: Consultation — Consultations at a specialist surgical nurse-led clinic
  Arms: Intervention

SUMMARY:
The main hypothesis is that a nurse-led education provided to patients who received endovascular treatment due to enlarged abdominal aorta would present a difference in perceived health, quality of life and sexual health.

DETAILED DESCRIPTION:
A longitudinal, prospective single-centre randomized control trial to evaluate the effects of a nurse-led educational intervention for patients undergoing endovascular intervention for abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* patients who received endovascular treatment for abdominal aortic aneurysm.
* patients who could understand and communicate in Swedish.

Exclusion Criteria:

* cognitive impairment or language impairment that prevents communication and informed consent.
* patients who did not receive endovascular treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Health Education Impact Questionnaire (HeiQ) | from enrollment to 12 month after enrollment
  A generic instrument (40 items), that measures health effects after education.
  The instrument consists of eight scales that measure different perceived health-related aspects:
  1. health directed activities, 2. positive and active engagement in life, 3. emotional distress, 4. self-monitoring and insight, 5. Constructive attitudes and approaches, 6. skills and technique acquisition, 7. social integration and support, and 8. health service navigation.
  The response options for each item are scored 1-4: "strongly disagree," "disagree," "agree" and "strongly agree."
  The HeiQ-scales are scored by summarizing within scale item scores, followed by dividing the sum with the number of scale items. A higher number represents better outcomes in all scales except for the emotional distress scale, where a higher score represents worse outcome.
Male Sexual Function-4 Questionnaire | from enrollment to 12 month after enrollment
  Questionnaire consisting of four items designed to asses aspects of sexual function, as well as perception of overall sexual quality of life.
  The four items include interest in sex, achieving orgasm, quality of erection, and achieving ejaculation. Each item is scored on a six-point Likert scale ranging from 0 to 5. The raw scores are linearly transformed to a global sex life index ranging from 0 to 100, where a lower score indicates better preserved sexual function.
  For female participants, four specific items related to female sexual function were used, based on MSF-4 and derived from a previous study that investigated female patients undergoing colorectal surgery; first two items were interest in sex and achieving orgasm and both used a six-point Likert scale ranging from 0 to 5 where a lower score indicates better outcome. The second two items were problems with insufficient vaginal moisture and changes in the vaginal sense postoperatively, both items used binary yes/no answers.

SECONDARY OUTCOMES:
EuroQol Five Dimension (EQ-5D-3L) | from enrollment to 12 month after enrollment
  standardized instrument designed to measure health outcomes that also has been commonly utilized in health economic analysis.
  An overall classification of perceived health is measured with a visual analog scale where 0 represents the worst possible imaginable health and 100 represents the best possible imaginable health. Health is further classified in five different dimensions: 1. mobility, 2. self-care, 3. daily activities, 4. pain/discomfort, and 5. depression/anxiety. These dimensions can be graded differently depending on what iteration of the instrument is being used. The present study used the three-scale step level version (EQ-5D-3L), with the alternatives "no problems," "some/moderate problems," and "extreme problems" for each dimension.
Complementary questions for the intervention | from enrollment to 12 month after enrollment
  Four complementary items were used to further evaluate the effects of the intervention in the form of visual analog scales: 1. degree of perceived understanding of the diagnosis (1= not at all and 100 = understands completely), 2. degree of perceived understanding of the purpose of postoperative medical imaging examinations (1 = not at all and 100 = understands completely), 3. degree of desire for additional information regarding their disease (0 = no, it is enough and 100 = yes, much more), 4. degree of perceived concern about treated AAA (0 = never and 100 = all the time).
Complementary questions for sexual function | from enrollment to 12 month after enrollment
  Three complementary content-specific items were added to investigate specific contextual aspects not covered by the MSF-4 questionnaire as follows: one question if the participants had received information regarding potential procedure-related effects on sexual health and function (with a binary yes/no answer), one question about the perceived satisfaction with the provided information (with a binary yes/no answer), and one question about experiencing concern during sexual activity (with a binary yes/no answer).
Laboratory analysis - Cholesterol | from enrollment to 12 month after enrollment
  blood analysis in mmol/L
Laboratory analysis - Triglycerids | from enrollment to 12 month after enrollment
  blood analysis in mmol/L
Laboratory analysis - High density lipoprotein (HDL) | from enrollment to 12 month after enrollment
  blood analysis in mmol/L
Laboratory analysis - Low density lipoprotein (LDL) | from enrollment to 12 month after enrollment
  blood analysis in mmol/L
Laboratory analysis - Plasma glucose | from enrollment to 12 month after enrollment
  blood analysis in mmol/L
Systolic blood pressure | from enrollment to 12 month after enrollment
  measured in mmHg
Diastolic blood pressure | from enrollment to 12 month after enrollment
  measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Monica Pettersson, Professor, Principal Investigator — Göteborg University